CLINICAL TRIAL: NCT00734188
Title: A Multi-Center, Open-Label, Phase I, Dose-Escalation and Safety Study of 188Re-PTI-6D2 in Patients With Metastatic Melanoma
Brief Title: Dose Escalation and Safety Study of 188Re-PTI-6D2 in Patients With Metastatic Melanoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pain Therapeutics (Industry)
Responsible Party: Eithan Galun, M.D., Hadassah Hebrew University Hospital
Organization: PainT (Unknown)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PTI-6D2-B
Record Dates: First submitted 2008-08-12; First posted 2008-08-14 (Estimated); Last update posted 2011-07-14 (Estimated); Status verified 2011-07

CONDITIONS: Metastatic Melanoma
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: PTI-6D2 — monoclonal antibody

SUMMARY:
This is an open-label, dose-escalation study to determine the safety, maximum tolerated dose (MTD) and dose-limiting toxicities (DLT) of 188Re-PTI-6D2 in patients with metastatic melanoma.

DETAILED DESCRIPTION:
Patients with confirmed Stage III (unresectable) or Stage IV melanoma who meet all eligibility criteria will undergo thorough physical examination and baseline tumor imaging to document baseline tumor measurements. Patients will be allowed to check in to the study center either the evening prior to dosing (Study Day 0) or the day of dosing (Study Day 1) based upon the principal investigators (PIs) discretion. All patients will be dosed and monitored as inpatients during the study.

Patients will receive an intravenous (IV) infusion of 188Re-PTI-6D2. Patients will undergo serial gamma scans at specified time points. Blood samples will be obtained prior to dosing and at specified intervals for PK measurements of the mAb as well as for measurement of serum radioactivity. Urine will be collected to measure excreted radioactivity. Patients will be closely monitored for safety throughout the duration of the study. Patients will remain at the study center for 48-72 hours after infusion of the radiolabeled dose to allow adequate time for post-treatment safety observation and rhenium decay. No investigational or commercial agents or therapies other than the study agent may be administered with the intent to treat the patient's malignancy during the inpatient treatment period.

After three evaluable patients have been followed for a minimum of 2-6 weeks after 188Re-PTI-6D2 infusion, the Principal Investigator and the PTI Medical Monitor will review safety data for patients at the current dose level. If there is no evidence of a dose-limiting toxicity, the dose of 188Re-PTI-6D2 will be escalated for the next cohort of patients. Dose escalation of 188Re-PTI-6D2 will occur according to the following titration scheme:

Level 1 = 20-30 mCi 188Re-PTI-6D2 / 10 - 50 mg of antibody

Level 2 = 40-60 mCi 188Re-PTI-6D2 / 10 - 50 mg of antibody

Level 3 = 75-100 mCi 188Re-PTI-6D2 / 50 - 100 mg of antibody

Level 4 = 125-150 mCi 188Re-PTI-6D2 / 50 - 100 mg of antibody

Level 5 = 175-200 mCi 188Re-PTI-6D2 / 50 - 100 mg of antibody

Dose-limiting toxicity will be defined as the following: Grade 4 hematological toxicity; ≥ Grade 3 non-hematological toxicity; or any adverse event that results in permanent discontinuation of the infusion. If at any time Grade 5 toxicity is observed, accrual will be suspended until further review. If 0 out of 3 patients experience DLT, the next cohort of 3 patients will be enrolled at the next dose level. If 1 out of 3 patients experience a dose-limiting toxicity, an additional three evaluable patients will be enrolled at the current dose level.

Dose escalation occurs until the maximum tolerated dose is determined. The MTD is defined as the dose preceding the dose at which 2 of 3 or 2 of 6 patients experience DLT.

Safety will be evaluated by vital signs (blood pressure, heart rate, respiratory rate and temperature), physical examinations, electrocardiograms (EKGs), clinical laboratory tests and adverse event monitoring. Laboratory studies will include hematology, chemistry and urinalysis at baseline, at the end of the inpatient treatment period, and at 2 weeks and 6 weeks after the infusion of the 188Re-PTI-6D2 dose. If hematological recovery has not occurred by week 6, patients will follow-up monthly until hematological recovery. In addition, thyroid function tests will be performed at baseline and at 6 weeks after infusion; then monthly until recovery (if has not occurred). Human anti-murine antibodies (HAMA) will be measured at baseline, 2 weeks, and 6 weeks after infusion .

Biodistribution of 188Re-PTI-6D2 will be evaluated by whole body imaging with a gamma camera immediately after infusion (0 - 2 hrs.), at 2.5 - 5 hours, at 6 - 8 hours, and 24 hours post-infusion. Whole body imaging at 48 and 72 hours post-infusion may be conducted at the discretion of the PI. Urine will be collected to measure cumulative radioactivity excretion up to 48-72 hours post-infusion (depending on the hospital discharge date). Pharmacokinetics of the mAb and radioactivity will be determined from blood samples taken through 48-72 hours post-infusion (depending on the hospital discharge date). Dosimetry calculations will be performed to determine estimated absorbed radiation doses to critical organs and to tumor.

Patients will be discharged from the study unit 48-72 hours after infusion with 188Re-PTI-6D2 or later as determined by the Investigator's clinical judgment. Patients will be required to return for post-treatment follow-up visits approximately 2 and 6 weeks (± two days) after infusion for safety monitoring. Ongoing follow-up visits will continue until disease progression every 4 weeks. Tumor measurements will be performed at baseline, and all follow-up visits to assess for tumor response. Patients with unacceptable adverse events will have events followed until resolution.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or clinically confirmed malignant melanoma of one of the following stages (according to 2002 American Joint Committee on Cancer criteria: Appendix C): Unresectable Stage III disease or Stage IV disease
* Patients must have measurable disease as defined by at least one target lesion ≥ 10 mm by spiral CT scan or ≥ 20 mm by conventional techniques
* Males or females ≥ 18 years of age
* Karnofsky performance status ≥ 60% (see Appendix D)
* Life expectancy of greater than three months
* Failure to respond to other therapy
* At least 4 weeks since prior chemotherapy or radiation therapy and at least one week since IL-2 therapy
* Patients must not have significant organ and marrow dysfunction as defined by the following Screening laboratory values: Leukocytes ≥ 3,000/mcL; Absolute neutrophil count ≥ 1,500/mcL; Platelets ≥ 50,000/mcL; Total bilirubin ≤ 2.0 × upper limit of normal(ULN); AST(SGOT)/ALT(SGPT) ≤ 3 × ULN or ≤ 6 × ULN if liver metastases present; Creatinine ≤ 2.0 or creatinine clearance ≥ 60 mL/min/1.73 m2 if creatinine > 2.0
* Patients must have negative screening human anti-murine antibodies (HAMA).
* Females who are postmenopausal, physically incapable of childbearing, or practicing an acceptable method of birth control. Acceptable methods of birth control include surgical sterilization, hormonal contraceptives, or double-barrier methods (condom or diaphragm with a spermicidal agent or IUD). If practicing an acceptable method of birth control, a negative urine pregnancy test result has been obtained at the Screening Visit
* Patients must be able to understand study procedures and must sign a written informed consent form prior to entering the study
* Patients must agree to comply with all treatment procedures and be willing and able to remain at the study site unit for no less than 48 hours after infusion with 188Re-PTI-6D2 or later as determined by the Investigator's clinical judgment

Exclusion Criteria:

* Patients who have had chemotherapy or radiotherapy within 4 weeks (IL-2 therapy within one week) prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier
* Patients who have participated in another investigational drug trial or therapeutic trial within 30 days of the Screening Visit
* Patients with brain metastases (must be confirmed by contrast-enhanced MRI within 4 weeks of study entry - a CT scan may be substituted for patients who cannot tolerate the MRI procedure)
* Patients with any ocular disease that, in the opinion of the PI, could lead to an impaired blood-retinal brain barrier: e.g. severe retinal detachment, ocular melanoma or other ocular neoplastic process, or ocular inflammatory disease
* Patients with a prior parenteral exposure to murine proteins or a history of allergy or hypersensitivity to investigational or approved antibodies
* HIV-positive patients on combination antiretroviral therapy are ineligible because of increased risk of lethal infections secondary to marrow-suppressive therapy
* Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Patients who are pregnant or breast-feeding
* Patients who are unwilling to reside in the study unit for a minimum of 48 hours after infusion with 188Re-PTI-6D2 or later as determined by the Investigator's clinical judgment, or to cooperate fully with the investigator or site personnel

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 2009-01; Primary Completion 2010-03 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
To determine the maximum tolerated dose (MTD) of 188Re-PTI-6D2 in patients with metastatic melanoma | Daily/Weekly/Monthy

SECONDARY OUTCOMES:
to determine safety and tolerability; dose-limiting toxicities; evaluate the anti-tumor activity; to evaluate the HAMA response; and, to further characterize the pharmacokinetics, biodistribution, and dosimetry of 188Re-PTI-6D2 | Daily/Weekly/Monthly

CONTACTS AND LOCATIONS:
Overall Officials: Eithan Galun, M.D., Principal Investigator — Hadassah Hebrew University Hospital
Locations (1):
- Hadassah Hebrew University Hospital, Jerusalem, Israel